CLINICAL TRIAL: NCT06637865
Title: A Placebo-controlled, Double-blind Phase I Study in Healthy Volunteers With IMP761, a LAG-3 Agonist Antibody
Brief Title: A First-in-human Study of the Safety of an Immunosuppressive Antibody (IMP761) in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IMP761-P001; 2024-510761-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — keyhole-limpet hemocyanin

STUDY DESIGN:
Intervention Model Description: There will be 10 cohorts in total: 8 single dose cohorts and 2 multiple dose cohorts
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Single ascending dose IMP761 Part A (Experimental): Randomized in 3:2 (IMP761:placebo) Cohort 1: 5 subjects
  Interventions: Drug: IMP761
- Single ascending dose Placebo Part A (Placebo Comparator): Randomized in 3:2 (IMP761:placebo) Cohort 1: 5 subjects
  Interventions: Drug: Placebo
- Single ascending dose IMP761 Part B KLH challenge (Experimental): Randomized in 4:1 (IMP761:placebo). KLH immunization followed by IMP761 on Day 1 and dermal rechallenge on day 2 (Cohorts 2-3) or on days 2, 9 and 23 (Cohorts 4-8)
  Cohort 2: 5 subjects; Cohort 3: 5 subjects; Cohort 4: 10 subjects; Cohort 5: 10 subjects; Cohort 6: 10 subjects; Cohort 7: 10 subjects; Cohort 8: 10 subjects
  Interventions: Drug: IMP761; Other: keyhole limpet haemocyanin (KLH)
- Single ascending dose Placebo Part B KLH challenge (Placebo Comparator): Randomized in 4:1 (IMP761:placebo). KLH immunization followed by placebo on Day 1 and dermal rechallenge on day 2 (Cohorts 2-3) or on days 2, 9 and 23 (Cohorts 4-8)
  Cohort 2: 5 subjects; Cohort 3: 5 subjects; Cohort 4: 10 subjects; Cohort 5: 10 subjects; Cohort 6: 10 subjects; Cohort 7: 10 subjects; Cohort 8: 10 subjects
  Interventions: Drug: Placebo; Other: keyhole limpet haemocyanin (KLH)
- Multiple ascending dose IMP761 Part C (Experimental): Randomized 5:2 (IMP761:placebo) every 28 days, 3 times. MAD Cohort 1: 7 subjects; MAD Cohort 2: 7 subjects
  Interventions: Drug: IMP761
- Multiple dose placebo Part C (Placebo Comparator): Randomized 5:2 (IMP761:placebo) every 28 days, 3 times. MAD Cohort 1: 7 subjects; MAD Cohort 2: 7 subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMP761 — intravenous
  Arms: Multiple ascending dose IMP761 Part C; Single ascending dose IMP761 Part A; Single ascending dose IMP761 Part B KLH challenge
Drug: Placebo — intravenous
  Arms: Multiple dose placebo Part C; Single ascending dose Placebo Part A; Single ascending dose Placebo Part B KLH challenge
Other: keyhole limpet haemocyanin (KLH) — intramuscular immunization and intradermal challenge
  Arms: Single ascending dose IMP761 Part B KLH challenge; Single ascending dose Placebo Part B KLH challenge

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of single and multiple doses of IMP761 in healthy female and male volunteers aged 18-55 with no history of disease affecting the immune system or recent use of medication with effects on the immune system.

The main question it aims to answer is:

- if IMP761 is safe and tolerable as determined by assessing vital signs, emerging (serious) adverse events, electrocardiography, and clinical laboratory tests.

Researchers will compare IMP761 to a placebo (a look-alike substance that contains no drug) to see if single and multiple doses of IMP761 are safe and tolerable in healthy volunteers. Part B of the study also investigates the effect of IMP761 on the inhibition of the keyhole limpet haemocyanin (KLH) driven immune response compared with placebo.

Participants will:

* receive IMP761 or a matching placebo intravenously once in single dose (part A and B) and three times in multiple dose (part C) during a 4 day in clinic stay with 4-8 following visits.
* receive KLH challenge
* be monitored for up to 103 days after the first dose.

DETAILED DESCRIPTION:
This is a first in human, randomized, prospective, single centre, double blind, placebo-controlled study in healthy volunteers. It consists of three separate parts (Part A, B and C) with different study designs.

The main objective is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending dose (SAD) (Part A and B) and multiple ascending doses (MAD) (Part C) of IMP761 as assessed by:

* Vital signs
* Treatment-emergent (serious) adverse events ((S)AEs)
* Electrocardiography.
* Clinical laboratory tests
* Laser speckle contrast imaging (LSCI)
* Multispectral skin imaging

Part A: SAD study in healthy subjects (cohort 1, 5 subjects) Cohort 1: 5 subjects, single i.v. dose of IMP761 or placebo (3:2). The first 2 subjects will receive IMP761 or placebo (1:1) as sentinel dosing, while the following 3 subjects will receive IMP761 or placebo (2:1).

Part B: SAD study in healthy subjects, KLH challenge (cohort 2-8, 60 subjects) Cohort 2-3: 5 subjects, single i.v. dose of IMP761or placebo (4:1). Cohort 4-8: 10 subjects, single i.v. dose of IMP761 or placebo (8:2).

Part C: MAD study in healthy subjects (MAD cohort 1-2, 14 subjects) MAD Cohort 1-2: 7 subjects, multiple (three i.v. doses of IMP761 or placebo (5:2). Investigational Medicinal Product (IMP)/placebo administration every 28 days; dose selection to be based on observed pharmacodynamic effects in part B.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and willing and able to comply with the study protocol;
2. Healthy men or women, 18 to 55 years of age (inclusive) at screening. The health status is verified by absence of evidence of any clinically significant active or uncontrolled chronic disease following a detailed medical history, a complete physical examination including vital signs, laboratory measurements, and 12-lead electrocardiogram (ECG);
3. Female subjects agree to use effective contraception for the duration of their participation in the study and until 186 days after End of Study (EOS).
4. Male volunteers agree to use barrier protection when they engage in sexual relations with women of child-bearing potential (WOCBP) or lactating women for the duration of their participation in the study and until 96 days after EOS.
5. Body mass index (BMI) between 18 and 32 kg/m2, inclusive, and with a minimum bodyweight of 50 kg;
6. Fitzpatrick skin type I-III (cohorts 2-5 only);
7. Has the ability to communicate well with the Investigator in Dutch language and willing to comply with the study restrictions.
8. Has the intention to be reachable by mobile phone or e-mail during the whole study period.

Exclusion Criteria:

1. Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator (following a detailed medical history, physical examination, vital signs (systolic and diastolic blood pressure, pulse rate, body temperature) and 12-lead electrocardiogram (ECG)). Minor deviations from the normal range may be accepted, if judged by the Investigator to have no clinical relevance;
2. Clinically significant abnormalities, as judged by the Investigator, in laboratory test results (including haematology panel, chemistry panel and urinalysis). In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility. A rescreen will be allowed based on judgement of the investigator;
3. Positive immunodeficiency virus (HIV1, HIV2) antigen or antibody, Hepatitis B surface antigen (HBsAg), Hepatitis B Virus antibody (HBV Ab), Hepatitis C antibody (HCV Ab), (latent) Tuberculosis at screening;
4. Any disease associated with immune system impairment, including immune mediated diseases, transplantation patients and any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug or multiple drug allergies (non-active hay fever is acceptable);
5. Use of any medications (prescription or over-the-counter [OTC]), within 21 days prior to dosing with Investigational Medicinal Product (IMP), or less than 5 half-lives (whichever is longer). An exception is made for paracetamol (up to 4 g/day).
6. Use of vitamin, mineral, herbal and dietary supplements within 7 days prior to study drug administration, which are deemed clinically significant by the investigator.
7. Use of immunosuppressive or immunomodulatory medication within 30 days prior to dosing with IMP or planned to use immunosuppressive or immunomodulatory medication during the course of the study.
8. Any vaccination within 30 days prior to dosing with IMP or planned during the course of the study or within 90 days after the last dose of IMP.
9. Use of antibiotic therapy within 90 days prior to dosing with IMP or planned to use during the course of the study.
10. Subject is unable to abstain from travelling to areas with high endemic rates of infectious diseases from study entry until 90 days after the last dose of IMP
11. Alcohol will not be allowed from at least 24 hours before screening and each scheduled visit. At other times during the course of the study no more than 2 units of alcohol per day will be allowed.
12. If a woman, pregnant, or breast-feeding, or planning to become pregnant during the study.
13. Have any current and/or recurrent clinically significant skin condition at the dermal challenge area (i.e. atopic dermatitis), including tattoos.
14. Any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinically relevant abnormalities in vital signs | From screening to the follow up visit after last treatment (up to 143 days)
Frequency of adverse events (AEs) | From administration to the follow up visit after last treatment (up to 103 days)
Duration of adverse events (AEs) | From administration to the follow up visit after last treatment (up to 103 days)
Severity of adverse events (AEs) | From administration to the follow up visit after last treatment (up to 103 days)
Occurrence of clinically relevant abnormalities in electrocardiography | From screening to the follow up visit after last treatment (up to 143 days)
Occurrence of clinically relevant abnormalities in safety laboratory assessments | From screening to the follow up visit after last treatment (up to 143 days)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter: Maximum Serum Concentration (Cmax) (Part B and C) | Up to 86 days
PK parameter: Timepoint of Maximum Serum Concentration (tmax) (Part B and C) | Up to 86 days
PK parameter: Minimum Serum concentration (Cmin) (Part B and C) | Up to 86 days
PK parameter: Area Under the Curve (AUC) (Part B and C) | Up to 86 days
PK parameter: systemic clearance (CL) (Part B and C) | Up to 86 days
PK parameter: Apparent volume of distribution at steady state (Vss) (Part B and C) | Up to 86 days
PK parameter: Apparent volume of distribution at terminal state (Vz) (Part B and C) | Up to 86 days
PK parameter: elimination half-life (t1/2) (Part B and C) | Up to 86 days
PK Parameter: Trough Concentration (Ctrough ) (Part C) | Up to 86 days
PK Parameter: Peak to trough ratio (PTR) (Part C) | Up to 86 days

OTHER OUTCOMES:
Pharmacodynamic (PD) parameter: Changes of erythema severity by multispectral skin imaging (Part B) | Day 2, 3, 9, 10, 23 and 24
PD parameter: Changes of erythema shape by multispectral skin imaging (Part B) | Day 2, 3, 9, 10, 23 and 24
PD parameter: Cutaneous microcirculation assessed using laser speckle contrast imaging (LSCI) (Part B) | Day 2, 3, 9, 10, 23 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- CHDR, Leiden, Netherlands